CLINICAL TRIAL: NCT03884413
Title: FErtility, PrEgnancy, contRaceptIon After Breast Cancer in France: the FEERIC Study
Brief Title: FErtility, PrEgnancy, contRaceptIon After Breast Cancer in France
Acronym: FEERIC
Status: Completed | Type: Observational
Sponsor: Institut Curie (Other)
Collaborators: seintinelles network (Unknown)
Responsible Party: Sponsor
Other Study IDs: IC 2016-07
Record Dates: First submitted 2018-11-02; First posted 2019-03-21 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2018-11

CONDITIONS: Breast Cancer Female
Keywords: breast cancer survivors,; spontaneous fertility rates,; pregnancy,; birth rate,; chemotherapy-induced infertility
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Breast cancer survivors: Study of spontaneous fertility outcomes following breast cancer history
  Interventions: Other: questionnaires
- Control group: Study of spontaneous fertility outcomes in healthy volonteers population
  Interventions: Other: questionnaires

INTERVENTIONS:
Other: questionnaires — Longitudinal observational study. Collection of health data using self-administered questionnaires online.

SUMMARY:
FErtility, PrEgnancy, contRaceptIon after breast Cancer in France

DETAILED DESCRIPTION:
Breast cancer is the most common cancer among women. With the increase of the survival rates, a growing attention is paid to the side effects of the treatments, particularly chemotherapy-induced infertility.

The FEERIC study will give insights into spontaneous fertility outcomes following breast cancer in comparison with a control cohort and will provide data to help patients counselling towards spontaneous fertility rates following breast cancer. It will also provide data on contraceptive prevalence and unintended pregnancy rates in French breast cancer survivors. Reasons for unmet need for family planning will be deciphered, in order to point out pitfalls (lack of patient's information or orientation/ignorance of contraception methods available/topic insufficiently or not discussed with the physician/ lack of family planning offer etc…); and target the appropriate actions to lead (oncologist and oncology nurses education/ dedicated consultations in breast cancer centers/etc…).

ELIGIBILITY:
Inclusion Criteria:

* females aged from 18 to 43 at inclusion
* previous diagnosis of breast cancer and time from diagnosis comprised between one and five years or women free from breast cancer or other malignancy (healthy volunteers) .

Exclusion Criteria:

* hysterectomy and/or bilateral oophorectomy and/or bilateral salpingectomy
* healthy volonteer with history of malignant disease.

Ages: 18 Years to 43 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women with previous diagnosis of breast cancer and time from diagnosis comprised between one and five years
Sampling Method: Non-Probability Sample
Enrollment: 517 (Actual)
Dates: Start 2018-03-08 (Actual); Primary Completion 2021-03-08 (Actual); Study Completion 2022-03-08 (Actual)

PRIMARY OUTCOMES:
Spontaneous pregnancies between cases and controls | 3 years
  Odds ratio between the spontaneous pregnancies between cases and controls, for women with a desire to become pregnant and trying to get pregnant.

SECONDARY OUTCOMES:
Time to spontaneous pregnancy | 3 years
  Time to spontaneous pregnancy after breast cancer diagnosis, for women with a desire to become pregnant and trying to get pregnant.
Contraceptive prevalence | 3 years
  Contraceptive use, defined as the percentage of women reporting use of a contraceptive method.
Rate of women considered with risk of unintended pregnancy | 3 years
  An unwanted pregnancy is defined as unwanted at the time of conception. Women are classified as at risk of unwanted pregnancy if they report having had unprotected sex without a desire to become pregnant in the previous four months.
Percentage of live births obtained by medically assisted procreation procedures | 3 years
  Percentages live births obtained by ARTs procédures, that include in vitro fertilization (IVF) and embryo transfer (ET), intracytoplasmic sperm injection (ICSI) and ovarian stimulation with exogenous gonadotropins.

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Sophie HAMY-PETIT, MD, Principal Investigator — Institut Curie
Locations (1):
- Seintinelles.Com, Paris, France

REFERENCES:
- [Result] Mangiardi-Veltin M, Sebbag C, Rousset-Jablonski C, Ray-Coquard I, Berkach C, Laot L, Wang Y, Abdennebi I, Labrosse J, Sautter C, Toussaint A, Sablone L, Laas E, Khallouch S, Coussy F, Santulli P, Chapron C, Bobrie A, Jacot W, Sella N, Dumas E, Senechal-Davin C, Espie M, Giacchetti S, Maitrot L, Plu-Bureau G, Coutant C, Guerin J, Asselain B, Fumoleau P, Rodrigues M, Decanter C, Mailliez A, Delrieu L, Lemoine A, Jouannaud C, Houdre D, Reyal F, Hamy AS; Seintinelles Research Network. Pregnancy, fertility concerns and fertility preservation procedures in a national study of French breast cancer survivors. Reprod Biomed Online. 2022 Jun;44(6):1031-1044. doi: 10.1016/j.rbmo.2021.12.019. Epub 2022 Jan 19. PMID 35525718